CLINICAL TRIAL: NCT03617367
Title: A Phase 3, Open-Label, Multi-Center Trial to Evaluate the Long-Term Safety and Efficacy of Repeat Treatments of DaxibotulinumtoxinA for Injection in Adults With Isolated Cervical Dystonia (ASPEN-OLS)
Brief Title: Long-Term Safety and Efficacy of Repeat Treatments of DaxibotulinumtoxinA for Injection in Adults With Isolated Cervical Dystonia (ASPEN-OLS)
Acronym: ASPEN-OLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1720304
Record Dates: First submitted 2018-07-12; First posted 2018-08-06 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Cervical Dystonia
Keywords: DAXI; Cervical Dystonia; TWSTRS; Toxin; multiple treatment
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, open-label, multi-center trial to evaluate the long-term safety, efficacy, and immunogenicity of up to four continuous treatment cycles of daxibotulinumtoxinA (DAXI) for injection with up to four different doses in adults with isolated cervical dystonia (CD).
Masking Description: not applicable (open label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- daxibotulinumtoxinA (DAXI) for injection (Experimental): DAXI for injection
  Interventions: Biological: daxibotulinumtoxinA for injection

INTERVENTIONS:
Biological: daxibotulinumtoxinA for injection — DaxibotulinumtoxinA for injection is a sterile, white to off-white lyophilized product containing the active ingredient, daxibotulinumtoxinA, and inactive ingredients to be reconstituted with sterile, non-preserved, 0.9% sodium chloride solution saline.

SUMMARY:
Phase 3, open-label, multi-center trial to evaluate the long-term safety, efficacy, and immunogenicity of up to four continuous treatment cycles of daxibotulinumtoxinA (DAXI) for injection.

DETAILED DESCRIPTION:
Approximately 350 adult subjects will be recruited from approximately 80 study centers in the United States, Canada, and Europe who were enrolled in the ASPEN-1 Study Protocol 1720302 and de novo subjects (not previously enrolled in ASPEN-1 Study Protocol 1720302) will be treated with up to 4 different doses of daxibotulinumtoxinA for injection.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for isolated CD (idiopathic; dystonic symptoms localized to the head, neck, shoulder areas) with at least moderate severity at Baseline (Day 1), defined as a TWSTRS-total score of at least 20, with at least 15 on the TWSTRS-Severity subscale, at least 3 on the TWSTRS-Disability subscale, and at least 1 on the TWSTRS-Pain subscale (minimum TWSTRS subscale criteria applicable only to subjects not previously enrolled in Study Protocol 1720302)
* Subjects who were previously enrolled in Study Protocol 1720302, and completed the study, including:

  * Those with no reduction or have an increase from baseline in the average TWSTRS-total score at Weeks 4 and 6 (i.e., no improvement or worsened disease status), and the investigator agreed that there was a need for retreatment based on the subject's symptoms and neurologic exam findings
  * Those who benefited from study treatment and completed follow-up study visits up to the time point of when their TWSTRS - total score reached/exceeded their target TWSTRS score
  * Those who benefited from study treatment but subsequently experienced significant recurrence of CD symptoms (e.g. pain) during the study before their TWSTRS-total score reached their target TWSTRS score and requested retreatment, which the investigator determined was warranted based on the subject's symptoms and neurologic exam findings
  * Those who completed study visits up to Week 36 and their TWSTRS-total score never reached their target TWSTRS score and they never requested another treatment. The investigator determined that these subjects can be followed in the OLS until their TWSTRS-total score is the same or higher than their target TWSTRS score or until they request retreatment, which the investigator determined is clinically indicated
* De novo subjects (not previously enrolled in Study Protocol 1720302):

  * Naïve to BoNT treatment
  * BoNT treatment-experienced; if previously treated with BoNTA, the subject must have demonstrated a clinically meaningful response to the last BoNTA treatment based on the clinical judgment of the investigator

Exclusion Criteria:

* Cervical dystonia attributable to an underlying etiology, (e.g., traumatic torticollis or tardive torticollis)
* Predominant retrocollis or anterocollis CD
* Significant dystonia in other body areas, or is currently being treated with botulinum toxin (BoNT) for dystonia in areas other than those associated with isolated CD
* Severe dysphagia (Grade 3 or 4 on the Dysphagia Severity Scale) at Screening or Baseline (prior to study treatment)
* Any neuromuscular neurological conditions that may place the subject at increased risk of morbidity with exposure to BoNT, including peripheral motor neuropathic diseases (e.g., amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis)
* Previous treatment with any BoNT product for any condition within the 14 weeks prior to Screening (applicable only to de novo subjects)
* Botulinum neurotoxin treatment-experienced subjects who had suboptimal or no treatment response to the most recent BoNTA injection for CD, as determined by the investigator; or history of primary or secondary non-response to BoNTA injections, known to have neutralizing antibodies to BoNTA; or have a history of botulinum toxin type B (rimabotulinumtoxinA [Myobloc/Neurobloc]) injection for CD due to non-response or suboptimal response to BoNTA (applicable only to de novo subjects)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Long Term Safety of patients determined by the incidence of treatment-emergent adverse events | Up to 52 Weeks
  Evaluation of adverse events and serious adverse events, from multiple continuous treatments of DAXI for injection, over the course of the study.

SECONDARY OUTCOMES:
The proportion of subjects with at least moderate improvement on the Clinician Global Impression of Change (CGIC) at Weeks 4 or 6 for Treatment Cycles 1, 2, 3, and 4 | Weeks 4 and 6 of treatment cycles 1, 2, 3, and 4 (12 - 52 weeks duration each)
  The CGIC is an investigator-reported assessment of the global clinical change in CD since study treatment administration. The CGIC uses a 7-point Likert scale ranging from +3 (very much improved) to -3 (very much worse), and will be assessed by the investigator at the Week 4 and Week 6 visits.
The average of the change from Baseline in the TWSTRS Total Score at Weeks 4 and 6 for Treatment Cycles 1, 2, 3, and 4 [Time Frame: Weeks 4 and 6 of treatment cycles 1, 2, 3, and 4 (12 - 52 weeks duration each)] | Weeks 4 and 6 of treatment cycles 1, 2, 3, and 4 (12 - 52 weeks duration each)
  The difference in TWSTRS-Total score between the Baseline and average of Weeks 4 and 6 for each treatment cycle will be determined for each subject. The TWSTRS is an assessment scale used to measure the impact of CD on subjects. TWSTRS-total score has a minimum score of 0 and a maximum score of 85, where higher scores represent worse outcomes. It is made up of the summation of 3 subscales: the Torticollis Severity Scale (minimum score of 0, maximum score of 35), the Disability Scale (minimum score of 0, maximum score of 30), and the Pain Scale (minimum score of 0, maximum score of 20).

CONTACTS AND LOCATIONS:
Locations (65):
- United States (37):
  - HOPE Research Institute, Phoenix, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - The Parkinsons and Movement Disorder Institute, Fountain Valley, California
  - Loma Linda University, Loma Linda, California
  - USC Keck School of Medicine, Los Angeles, California
  - Care Access Research LLC, Pasadena, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Infinity Clinical research, Hollywood, Florida
  - University of Miami, Miami, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas Institute of Research, Overland Park, Kansas
  - Michigan State University, East Lansing, Michigan
  - QUEST Research Institute, Farmington, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - St Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Movement Disorders Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Coastal Neurology, Port Royal, South Carolina
  - Intrafusion Research Network - Wesley Neurology Clinic, Cordova, Tennessee
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology. P.A., Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
- Neurologisches Studienzentrum Universitätsklinik für Neurologie Innsbruck, Innsbruck, Austria
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada
- Czechia (4):
  - Fakultní nemocnice Ostrava, Ostrava-Poruba
  - Nemocnice Pardubickeho kraje, a.s.; Pardubicka nemocnice, Pardubice
  - Neurologicka klinika 1. LF UK a VFN v Praze, Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- France (4):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU de Grenoble, Grenoble
  - Hôpital Roger Salengro, Lille
  - CHU Caremeau, Nîmes
- Germany (5):
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar der TUM, München
  - GFO Kliniken Troisdorf, Betriebsstätte St. Johannes Sieglar, Troisdorf
  - Universitätsklinikum Tübingen, Tübingen
- Poland (6):
  - Szpital sw. Wojciecha Podmiot Leczniczy Copernicus Sp. Z o.o., Gdansk
  - Marta Dagmara BANACH Marta Banach Specjalistyczny Gabinet Neurologiczny, Krakow
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Mazovian Brodno Hospital, Warsaw
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Burgos, Burgos
  - Hospital Universitario de La Princesa, Madrid
- United Kingdom (3):
  - Royal Devon and Exeter Foundation Trust Hospital, Exeter
  - The Walton Centre NHS Foundation Trust, Neuroscience Research Centre, Liverpool
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McAllister P, Patel AT, Banach M, Ellenbogen A, Slawek J, Paus S, Jinnah HA, Evidente V, Gross TM, Kazerooni R, Gallagher CJ, Hollander DA. Long-Term Safety and Efficacy of Repeat Treatments with DaxibotulinumtoxinA in Cervical Dystonia: Results from the ASPEN-Open-Label Study. Mov Disord Clin Pract. 2025 Nov;12(11):1764-1773. doi: 10.1002/mdc3.70104. Epub 2025 May 29. PMID 40439027